CLINICAL TRIAL: NCT06691191
Title: Switching From Dual Antiplatelet Therapy to Monotherapy With Potent P2Y12 Inhibitors: Pharmadodynamic Comparison Between Prasugrel and Ticagrelor Monotherapy. The Switching Antiplatelet -7 (SWAP-7) Study
Brief Title: Switching From Dual Antiplatelet Therapy to Monotherapy With Potent P2Y12 Inhibitors
Acronym: SWAP-7
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202401578
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; ticagrelor; prasugrel; bleeding; platelets
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Intervention Model Description: The proposed investigation will be a prospective, randomized, parallel-design, open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor monotherapy (Active Comparator): Ticagrelor 90 mg bid monotherapy for 21±7 days
  Interventions: Drug: Ticagrelor 90 mg
- Prasugrel monotherapy (Experimental): Prasugrel 10 mg qd for 21±7 days
  Interventions: Drug: Prasugrel 10 mg

INTERVENTIONS:
Drug: Ticagrelor 90 mg — After providing written informed consent, patients on DAPT meeting study entry criteria will stop aspirin and be randomly assigned in a 1:1 fashion using a computer-based randomization system to either: a) ticagrelor 90 mg bid monotherapy or b) prasugrel 10 mg qd monotherapy. Patients will continue the randomized treatment for 21±7 days.
  Other Names: Brilinta
  Arms: Ticagrelor monotherapy
Drug: Prasugrel 10 mg — After providing written informed consent, patients on DAPT meeting study entry criteria will stop aspirin and be randomly assigned in a 1:1 fashion using a computer-based randomization system to either: a) ticagrelor 90 mg bid monotherapy or b) prasugrel 10 mg qd monotherapy. Patients will continue the randomized treatment for 21±7 days.
  Other Names: Effient
  Arms: Prasugrel monotherapy

SUMMARY:
Ticagrelor currently represents the most tested and commonly used P2Y12 inhibitor monotherapy following percutaneous coronary intervention. The purpose of this study is to conduct a head-to-head comparison on the pharmacodynamic efficacy of ticagrelor-based and prasugrel-based single antiplatelet therapy. To determine if the PD profiles of ticagrelor- and prasugrel-based SAPT are comparable, we aim to conduct a non-inferiority study between the two strategies.

DETAILED DESCRIPTION:
A strategy of P2Y12 monotherapy after 1-3 months of dual antiplatelet therapy (DAPT) is associated with a substantial reduction in bleeding events without an increase in atherothrombotic events, including in patients with acute coronary syndrome (ACS). However, different P2Y12 inhibitors vary in safety and efficacy profiles in the setting of single antiplatelet therapy (SAPT). In the TICO (Ticagrelor Monotherapy After 3 Months in the Patients Treated With New Generation Sirolimus-eluting Stent for Acute Coronary Syndrome) trial, DAPT discontinuation at 3 months with transition to ticagrelor monotherapy was superior to standard 12-month DAPT for 1-year net adverse cardiac events in ACS patients undergoing percutaneous coronary intervention (PCI). Similarly, the TWILIGHT (Ticagrelor with Aspirin or Alone in High-Risk Patients after Coronary Intervention) trial showed that in high-risk patients who have completed an initial 3-month course of DAPT following PCI, ticagrelor monotherapy reduced clinically meaningful bleeding events without increasing ischemic risk as compared with ticagrelor plus aspirin. In contrast, in STOPDAPT-2 ACS (Short and Optimal Duration of Dual Antiplatelet Therapy-2 Study for the Patients With ACS), discontinuation of DAPT at 1 to 2 months after ACS PCI with transition to clopidogrel monotherapy was not noninferior to 12-month DAPT with aspirin and clopidogrel for 1-year net adverse cardiac events, due to a numerical increase in atherothrombotic events despite reduction in bleeding events. These data suggest that potent P2Y12 inhibitors should be preferred over clopidogrel in the setting of early SAPT after PCI in high-risk patients.

The ISAR-REACT (Intracoronary Stenting and Antithrombotic Regimen: Rapid Early Action for Coronary Treatment) 5 trial showed that in ACS patients the incidence of major cardiovascular events was lower among those who received prasugrel than among those who received ticagrelor, and the incidence of major bleeding was not significantly different between the two groups. Based on these findings, European guidelines now suggest that prasugrel should be considered in preference to ticagrelor for ACS patients who proceed to PCI. Moreover, PD studies showed that, compared with ticagrelor, prasugrel provides similar or even superior platelet inhibition [16,17]. However, this clinical PD data is in the context of using prasugrel in the context of a DAPT regimen (i.e., in adjunct to aspirin) and data on the use of prasugrel-based SAPT following PCI are limited.

Overall, these observations as well as the lack of head-to-head comparisons on the clinical and PD efficacy of ticagrelor-based and prasugrel-based SAPT underscore the importance of conducting dedicated investigations to compare these approaches. To determine if the PD profiles of ticagrelor- and prasugrel-based SAPT are comparable, we aim to conduct a non-inferiority study between the two strategies. Such investigation may provide insights into the safety and efficacy of these strategies and set the foundation for larger-scale investigations assessing clinical outcomes.

ELIGIBILITY:
Inclusion criteria:

1. Patients on DAPT with aspirin plus prasugrel 10 mg or ticagrelor 90 mg bid as per standard of care at least 90 days after PCI.
2. Age between 18 and 75 years old
3. Able to provide written informed consent

Exclusion criteria:

1. Prior history of stent thrombosis
2. PCI within 90 days.
3. History of stroke/TIA
4. Age > 75 years old
5. Weight < 60 kg
6. History of intracranial hemorrhage
7. On treatment with any oral anticoagulant or chronic low-molecular-weight heparin (at venous thrombosis treatment, not for prophylaxis)
8. Patients with known coagulation disorders
9. Known severe hepatic impairment
10. Hypersensitivity to prasugrel or ticagrelor
11. Pregnant and breastfeeding persons [persons of childbearing age must use reliable birth control (i.e., oral contraceptives) while participating in the study]. If the potential subject is a person of childbearing potential, a pregnancy test will be done. If the subject is pregnant, participation in this study will end.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity measured by VerifyNow | 21±7 days
  The primary endpoint of the study is the comparison of P2Y12 reaction unites (PRU) levels determined by VerifyNow between prasugrel monotherapy and ticagrelor monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Franchi, MD, Principal Investigator — University of Florida College of Medicine Jacksonville
Locations (1):
- University of Florida Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No